**Study:** A Feasibility Study of Delivering Adolescent Nutrition Interventions Through School-Based Platforms in Ethiopia: A Cluster-Randomized Evaluation

Clinicaltrials.gov: NCT04121559

Document date: January 15, 2021

# ASSENT OF RESPONDENT (ADOLESCENT FEMALE AGED 10-14Y)

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention guidelines.

My name is <u>[NAME OF INTERVIEWER]</u>. I am a member of a survey team from Addis Continental Institute of Public Health (ACIPH), a research organization based in Addis Ababa. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive and Thrive program on adolescent health and nutrition in this area.

We want to talk with you about health and nutrition. We will also be asking you questions about your school attendance and experience. The information that you provide us will be used to improve the nutrition of adolescents in this community and across Ethiopia.

The interview may last for about two hours.

The information you will give us will not be disclosed to anyone. It will be kept strictly confidential.

There will be no cost to you other than your time. Your participation in the interview is voluntary. You have the right to not participate if you do not want to. You also have the right to refuse to answer specific questions or to stop this interview at any point during the interview. Not participating will not affect you or your family.

Your participation will be highly appreciated. The answers you give will help provide better information to policymakers and practitioners so that they can plan for better services that will respond to your needs.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the interview, or you can talk with:

Dr. Yemane Berhane

Director, Addis Continental Institute of Public Health Address: Yeka Sub City, Woreda 13, House No. B227 Tel: +251 116 390039 | Email: yemaneberhane@gmail.com-

Dr. Lieven Huybregts Research Fellow and IRB Chair International Food Policy Research Institute

Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

Tel: +1 202-862-6481 | Email: <a href="mailto:l.huybregts@cgiar.org">l.huybregts@cgiar.org</a>

The researcher read to me orally and explained the assent form. I understand that I am free to discontinue participation at any time if I so choose, and that the investigator will gladly answer any questions that arise.

| Do you agree to participate in this study? | No | 0 |
|--------------------------------------------|-----|---|
| | Yes | 1 |

| Interviewer's signature: | Date: | / | 1 | |
|--------------------------|-------|-----|-------|------|
| | | DAY | MONTH | YEAR |

# CONSENT OF RESPONDENT'S (ADOLESCENT FEMALE AGED 10-14Y) PARENT

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention guidelines.

My name is <u>[NAME OF INTERVIEWER]</u>. I am a member of a survey team from Addis Continental Institute of Public Health (ACIPH), a research organization based in Addis Ababa. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive and Thrive program on adolescent health and nutrition in this area.

We want to talk with your daughter about health and nutrition and also about her school attendance and experience. The information that she provides us will be used to improve the diet and nutrition of adolescents in this community and across Ethiopia.

We are requesting your permission for your daughter to be a participant in this study. The interview will last for about two hours. The information she provides us will be kept strictly confidential and will be used only for the study purposes.

There will be no cost to you or your daughter other than her time. Her participation in the interview is voluntary. She has the right to not participate if she does not want to. She will also have the right to refuse to answer specific questions or to stop the interview at any point during the interview. Not participating will not affect her or your family.

Your permission for your daughter's participation will be highly appreciated. The answers she gives will help provide better information to policymakers and practitioners so that they can plan for better services that will respond to adolescents' needs.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you and your daughter, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide your daughter with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you or your daughter have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the interview, or you can talk with:

Dr. Yemane Berhane

Director

Addis Continental Institute of Public Health

Address: Yeka Sub City, Woreda 13, House No. B227 Tel: +251 116 390039 | Email: yemaneberhane@gmail.com

Dr. Lieven Huybregts Research Fellow and IRB Chair International Food Policy Research Institute

Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

Tel: +1 202-862-6481 | Email: I.huybregts@cgiar.org

The researcher read to me orally and explained the consent form. I understand that I am free to discontinue my daughter's participation at any time if I so choose, and that the investigator will gladly answer any questions that arise.

| | Do you give permission for your daughter to participate in this study? | No 0<br>Yes 1 |
|---|---|---|
| Intervi | ewer's signature: | Date:///YEAR |

# CONSENT OF RESPONDENT (HEALTH EXTENSION WORKER)

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention guidelines.

My name is <u>[NAME OF INTERVIEWER]</u>. I am a member of a survey team from Addis Continental Institute of Public Health (ACIPH), a research organization based in Addis Ababa. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive and Thrive program on adolescent nutrition in this area.

We want to talk with you about the nutrition-related activities and services that you provide at primary schools and in the community. We will also be asking you questions about training and supervision that you received. The information that you provide us will be used to improve adolescent health and nutrition in this area and across Ethiopia.

The interview may last for about one hour.

The information you will give us will not be disclosed to anyone. It will be kept strictly confidential.

There will be no cost to you other than your time. Your participation in the interview is voluntary. You have the right to not participate if you do not want to. You also have the right to refuse to answer specific questions or to stop this interview at any point during the interview. Not participating will not affect you or your work.

Your participation will be highly appreciated. The answers you give will help provide better information to policymakers and practitioners so that they can plan for better services that will respond to your needs.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the interview, or you can talk with:

Dr. Yemane Berhane

Director, Addis Continental Institute of Public Health Address: Yeka Sub City, Woreda 13, House No. B227 Tel: +251 116 390039 | Email: yemaneberhane@gmail.com

Dr. Lieven Huybregts Research Fellow and IRB Chair International Food Policy Research Institute

Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

Tel: +1 202-862-6481 | Email: <a href="mailto:l.huybregts@cgiar.org">l.huybregts@cgiar.org</a>

The researcher read to me orally and explained the consent form. I understand that I am free to discontinue participation at any time if I so choose, and that the investigator will gladly answer any questions that arise.

| Do you agree to participate in this study? | No | 0 |
|--------------------------------------------|-----|---|
| | Yes | 1 |

| Interviewer's signature: | Date: | / | / | / |
|--------------------------|-------|-----|-------|------|
| | , | DAY | MONTH | YEAR |

# CONSENT OF RESPONDENT(S) (PARENT OF ADOLESCENT FEMALE AGED 10-14Y)

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention guidelines.

My name is <u>[NAME OF INTERVIEWER]</u>. I am a member of a survey team from Addis Continental Institute of Public Health (ACIPH), a research organization based in Addis Ababa. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive and Thrive program on adolescent health and nutrition in this area.

We want to talk with you about adolescent health and nutrition. We will also be asking you questions about your household. The information that you provide us will be used to improve the nutrition of adolescents in this community and across Ethiopia.

The interview may last for about one hour.

The information you will give us will not be disclosed to anyone. It will be kept strictly confidential.

There will be no cost to you other than your time. Your participation in the interview is voluntary. You have the right to not participate if you do not want to. You also have the right to refuse to answer specific questions or to stop this interview at any point during the interview. Not participating will not affect you or your family.

Your participation will be highly appreciated. The answers you give will help provide better information to policymakers and practitioners so that they can plan for better services that will respond to the needs of adolescents.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the interview, or you can talk with:

Dr. Yemane Berhane

Director, Addis Continental Institute of Public Health Address: Yeka Sub City, Woreda 13, House No. B227 Tel: +251 116 390039 | Email: yemaneberhane@gmail.com

Dr. Lieven Huybregts
Research Fellow and IRB Chair
International Food Policy Research Institute

Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

Tel: +1 202-862-6481 | Email: <a href="mailto:l.huybregts@cgiar.org">l.huybregts@cgiar.org</a>

The researcher read to me orally and explained the consent form. I understand that I am free to discontinue participation at any time if I so choose, and that the investigator will gladly answer any questions that arise.

| Mother: | |
|--------------------------------------------|---------------|
| Do you agree to participate in this study? | No 0<br>Yes 1 |
| Father: | |

| | Do you agree to participate in this study? | No<br>Yes | | . 0<br>1 |
|---|---|---|---|---|
| Intervie | ewer's signature: | Date: | / | / |
| | | | DAY M | ONTH |

# CONSENT OF RESPONDENT (SCHOOL TEACHER/PRINCIPAL)

Thank you for speaking with us today.

This interview will be held in accordance with COVID-19 prevention guidelines.

My name is <u>[NAME OF INTERVIEWER]</u>. I am a member of a survey team from Addis Continental Institute of Public Health (ACIPH), a research organization based in Addis Ababa. Together with the International Food Policy Research Institute (IFPRI), we are studying the Alive and Thrive program on adolescent nutrition in this area.

We want to talk with you about the activities provided at this school and in the community. We will also be asking you questions about nutrition-related activities and interventions that you conduct. The information that you provide us will be used to improve adolescent health and nutrition services in this area and across Ethiopia.

The interview may last for about one hour.

The information you will give us will not be disclosed to anyone. It will be kept strictly confidential.

There will be no cost to you other than your time. Your participation in the interview is voluntary. You have the right to not participate if you do not want to. You also have the right to refuse to answer specific questions or to stop this interview at any point during the interview. Not participating will not affect you or your work.

Your participation will be highly appreciated. The answers you give will help provide better information to policymakers and practitioners so that they can plan for better services that will respond to the needs of adolescents.

Contact with our survey team presents a risk of spreading COVID-19, an illness that can spread from person to person. To protect you, our survey team members will maintain two meters of distance, wear a mask, and wash or sanitize hands before and after the interview. We will also provide you with a mask. Each member of our survey team was checked for any symptoms of COVID-19 before starting work today. We ask that you let us know whether you have experienced any COVID-19 related symptoms today, so that additional safety measures can be applied if needed.

If you have any questions concerning the study, you may ask questions at any time before agreeing to participate or during the interview, or you can talk with:

Dr. Yemane Berhane

Director, Addis Continental Institute of Public Health Address: Yeka Sub City, Woreda 13, House No. B227

Tel: +1 202-862-6481 | Email: I.huybregts@cgiar.org

Tel: +251 116 390039 | Email: yemaneberhane@gmail.com-

Dr. Lieven Huybregts Research Fellow and IRB Chair International Food Policy Research Institute Address: 1201 Eye St. NW, Washington, DC 20005-3915 USA

The researcher read to me orally and explained the consent form. I understand that I am free to discontinue participation at any time if I so choose, and that the investigator will gladly answer any questions that arise.

| Do you agree to participate in this study? | No 0 |
|--------------------------------------------|-------|
| | Yes 1 |

| Interviewer's signature: | Date: | / | / | / |
|--------------------------|-------|-----|-------|------|
| | , | DAY | MONTH | YEAR |